CLINICAL TRIAL: NCT06269601
Title: The Reliability of the Upper Limb Rotation Test in Adolescent Male Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Birgül Dıngırdan, Master's degree, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: HÜ- FTR- BD- 02
Record Dates: First submitted 2024-02-02; First posted 2024-02-21 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Sports Physical Therapy
Keywords: Physical performance test; assessment; shoulder

STUDY DESIGN:
Intervention Model Description: 14-18 years basketball players
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- adolescent male basketball players (Other): 14-16 years adolescent male basketball players
  Interventions: Diagnostic Test: Upper Limb Rotation Test

INTERVENTIONS:
Diagnostic Test: Upper Limb Rotation Test — The athletes were instructed to perform a 90° abduction and 90° external rotation of the shoulder, accompanied by trunk rotation for a duration of 15 seconds. The number of repetitions was recorded. The tested side was the upper extremity in which the closed kinetic chain position was maintained. The test was repeated three times, and the average of the results was calculated.

SUMMARY:
The objective of the study is to examine the reliability of the Upper Limb Rotation Test in adolescent male basketball players aged between 14 and 16. According to the sample size calculation for the study, 51 athletes were included. The Upper Limb Rotation Test was administered to the athletes twice, with a one-week interval. The athlete was positioned in a plank stance with shoulder, elbow lateral epicondyle, greater trochanter, and ankle lateral malleolus making contact with the wall. The athletes were instructed to perform a 90° abduction and 90° external rotation of the shoulder, accompanied by trunk rotation for a duration of 15 seconds. The number of repetitions was recorded. The tested side was the upper extremity in which the closed kinetic chain position was maintained. The test was repeated three times, and the average of the results was calculated. The Upper Extremity Rotation Test is a reliable assessment tool for evaluating performance in adolescent basketball players aged 14-16, particularly in relation to shooting skills.

DETAILED DESCRIPTION:
The objective of the study is to examine the reliability of the Upper Limb Rotation Test in adolescent male basketball players aged between 14 and 16. According to the sample size calculation for the study, 51 athletes were included. The Upper Limb Rotation Test was administered to the athletes twice, with a one-week interval. The athlete was positioned in a plank stance with shoulder, elbow lateral epicondyle, greater trochanter, and ankle lateral malleolus making contact with the wall. The athletes were instructed to perform a 90° abduction and 90° external rotation of the shoulder, accompanied by trunk rotation for a duration of 15 seconds. The number of repetitions was recorded. The tested side was the upper extremity in which the closed kinetic chain position was maintained. The test was repeated three times, and the average of the results was calculated. The ICC (intraclass correlation coefficient) value, SEM (standard error of measurement), and MDC (minimal detectable change) values were calculated to assess the test-retest reliability of the evaluation tool. A low SEM value indicates higher reliability of measurements. The MDC value represents the smallest detectable change between two measurements. Differences below this value are considered practically undetectable or statistically insignificant.

ELIGIBILITY:
Inclusion Criteria:

* Male basketball players aged 14 to 18 years old.
* The athlete must have been engaged in basketball for a minimum of 3 years
* Athletes should be training at least three days per week.

Exclusion Criteria:

* The presence of coordination issues to an extent that hinders the compliance with the physiotherapist's instructions.
* Having undergone any orthopedic surgery in the upper extremities or spine within the last year.

Ages: 14 Years to 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 51 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-09-15 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
The Reliability of the Upper Limb Rotation Test | through study completion, an average of 1 year
  The Upper Limb Rotation Test was administered to the athletes twice with a one-week interval between the tests. The athlete was positioned in a plank position with shoulder, elbow lateral epicondyle, greater trochanter, and ankle lateral malleolus touching the wall. The athletes were instructed to perform a 90° shoulder abduction and 90° external rotation, along with a body rotation, for a duration of 15 seconds. The number of repetitions was recorded. The tested side involves the upper extremity where a closed kinetic chain position is maintained. The test was repeated three times, and the average of the results was calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Birgül Dıngırdan, Master, Study Chair — Hacettepe University; Volga Bayrakcı Tunay, Proffessor, Study Director — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gultekinler BD, Kaya BB, Gelen E, Tunay VB. The reliability of upper limb rotation test in adolescent male basketball players. BMC Sports Sci Med Rehabil. 2025 Nov 22;18(1):51. doi: 10.1186/s13102-025-01434-6. PMID 41275272